CLINICAL TRIAL: NCT01248416
Title: A Randomized Controlled Trial Of The Use Of Aromatase Inhibitors, Alone And In Combination With Growth Hormone In Adolescent Boys With Idiopathic Short Stature
Brief Title: Aromatase Inhibitors, Alone And In Combination With Growth Hormone In Adolescent Boys With Idiopathic Short Stature
Acronym: ThrasherAI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thrasher Research Fund (Other); Genentech, Inc. (Industry); Novartis (Industry); AstraZeneca (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, Chief, Division of Endocrinology, Diabetes & Metabolism, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180984
Record Dates: First submitted 2010-11-02; First posted 2010-11-25 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Idiopathic Short Stature
Keywords: Aromatase; Growth; Letrozole; Anastrozole; GH; Children; Puberty
MeSH Terms: interventions — Aromatase Inhibitors; Anastrozole; Letrozole; Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aromatase Inhibitor (Active Comparator): Anastrozole 1mg or Letrozole 2.5mg daily orally for 2 to 3 years
  Interventions: Drug: Aromatase Inhibitor
- Growth Hormone (Active Comparator): Somatropin 0.3mg/kg/week divided daily subcutaneously for 2 to 3 years
  Interventions: Drug: Growth Hormone
- Aromatase Inhibitor and Growth Hormone (Active Comparator): Anastrozole 1mg or Letrozole 2.5mg orally daily for 2 to 3 years and Somatropin 0.3mg/kg/week divided daily subcutaneously for 2 to 3 years
  Interventions: Drug: Aromatase Inhibitor; Drug: Growth Hormone; Drug: Aromatase Inhibitor and Growth Hormone

INTERVENTIONS:
Drug: Aromatase Inhibitor
  Other Names: Arimidex (Anastrozole); Femara (Letrozole)
  Arms: Aromatase Inhibitor; Aromatase Inhibitor and Growth Hormone
Drug: Growth Hormone
  Other Names: Nutropin (Somatropin); Genotropin (Somatropin)
  Arms: Aromatase Inhibitor and Growth Hormone; Growth Hormone
Drug: Aromatase Inhibitor and Growth Hormone
  Other Names: Arimidex (Anastrozole); Femara (Letrozole); Nutropin (Somatropin); Genotropin (Somatropin)
  Arms: Aromatase Inhibitor and Growth Hormone

SUMMARY:
When treating very short children in puberty we are time-limited, as sex hormones cause the growth plates to fuse and growth to end. Growth Hormone (GH), plus drugs that stop puberty, increase height potential, but leave children sexually infantile at a critical time in development. Human and animal data show that estrogen, in females and males, is a principal regulator of the fusion of the growth plate in puberty. Using aromatase inhibitors (AIs), which block testosterone to estrogen conversion, in boys with different growth disorders, we have shown that AIs may have beneficial effects enhancing height potential in growth-retarded males, without affecting their puberty. However, no direct comparison of the effect of AIs alone vs. conventional GH treatment has been done to date. This study will assess the effect of AIs alone, GH alone and combination treatment in enhancing height potential in adolescent boys with idiopathic short stature.

ELIGIBILITY:
Inclusion Criteria:

* Males: Ages: 12 - less than 18 years.
* Bone age less than 14 ½ years at study initiation.
* Presence of puberty.
* Idiopathic short stature will be defined as a short child equal or less than -2SD for height, with normal GH responses to stimuli (> or = 5ng/ml to at least 2 secretagogues) or a normal IGF-I and BP-3, normal body proportions and no other identifiable growth pathology.
* Accurate growth data for at least 6 months at baseline is available.

Exclusion Criteria:

* Chronic illnesses.
* Chronic use of glucocorticosteroids.
* Previous use of hormonal treatment with AIs, sex steroids or GH in the preceding 6 months.
* Birth weight small for gestational age (SGA).

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2010-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic Jacksonville
Locations (4):
- United States (3):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Nemours Children's Clinic- Jefferson, Philadelphia, Pennsylvania
- Veronica Mericq, MD, Santiago, Chile

REFERENCES:
- [Result] Mauras N, Ross JL, Gagliardi P, Yu YM, Hossain J, Permuy J, Damaso L, Merinbaum D, Singh RJ, Gaete X, Mericq V. Randomized Trial of Aromatase Inhibitors, Growth Hormone, or Combination in Pubertal Boys with Idiopathic, Short Stature. J Clin Endocrinol Metab. 2016 Dec;101(12):4984-4993. doi: 10.1210/jc.2016-2891. Epub 2016 Oct 6. PMID 27710241

RESULTS

PARTICIPANT FLOW:
Groups:
- Aromatase Inhibitor: Anastrozole 1mg or Letrozole 2.5mg daily orally for 2 to 3 years
  Aromatase Inhibitor
- Growth Hormone: Somatropin 0.3mg/kg/week divided daily subcutaneously for 2 to 3 years
  Growth Hormone
- Aromatase Inhibitor and Growth Hormone: Anastrozole 1mg or Letrozole 2.5mg orally daily for 2 to 3 years and Somatropin 0.3mg/kg/week divided daily subcutaneously for 2 to 3 years
  Aromatase Inhibitor
  Growth Hormone
  Aromatase Inhibitor and Growth Hormone
Period: Overall Study
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Started | 25 | 25 | 26
Completed | 21 | 25 | 25
Not Completed | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone | Total
Number analyzed (Participants) | 25 | 25 | 26 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.0) | 14.1 (1.2) | 14.0 (1.1) | 14.1 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 25 | 25 | 26 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Height
Description: Differences in height gains
Time Frame: 0 to 24 months
Population: Differences in height gains from 0 to 24 months; Of the 76 Subjects, 65 completed all procedures at 24 months.
Measure: Mean (Standard Error); unit: Centimeters
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 23
Centimeters | 14 (0.8) | 17.1 (0.9) | 18.9 (0.8)
Statistical Analysis 1: Comparison: Aromatase Inhibitor vs Growth Hormone vs Aromatase Inhibitor and Growth Hormone; Test type: Superiority; p < 0.006, ANCOVA

2. Primary Outcome: Change in Predicted Height
Description: Primary efficacy end point: change in predicted height (cm) from baseline at 24 months based on change in bone age (years)
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 23
centimeters | 0.5 (1.0) | 4.9 (0.9) | 7.4 (0.9)

3. Secondary Outcome: Change in Bone Density z Score Adjusted for Height
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months, however, 2 Subjects had a screw/pin in their leg/hip at the 24 month visit, and therefore, could not have a DEXA scan performed (N=63).
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 23
z-score | -1.061 (0.313) | -0.586 (0.244) | -0.605 (0.257)
Statistical Analysis 1: Comparison: Aromatase Inhibitor vs Growth Hormone vs Aromatase Inhibitor and Growth Hormone; Test type: Superiority; p = 0.906, ANOVA

4. Secondary Outcome: Change in Lean Body Mass
Time Frame: 0 to 24 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: kg
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 23 | 22
kg | 42.2 (1.6) | 42.0 (1.3) | 46.5 (1.2)
Statistical Analysis 1: Comparison: Aromatase Inhibitor vs Growth Hormone vs Aromatase Inhibitor and Growth Hormone; Test type: Superiority; p = 0.015, ANOVA

5. Secondary Outcome: Change in Body Mass Index
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 23
kg/m^2 | 2.5 (0.3) | 1.7 (0.4) | 2.5 (0.4)

6. Secondary Outcome: Change in IGF-I Concentrations
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months, however, 1 Subject, did not have IGF-1 results available for the 24 month visit (N=64).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 17 | 24 | 23
ng/mL | 158 (14) | 280 (16) | 303 (27)
Statistical Analysis 1: Comparison: Aromatase Inhibitor vs Growth Hormone; Test type: Superiority; p < 0.0001, ANOVA

7. Secondary Outcome: Change in Testosterone
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months.
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 23
ng/dL | 737 (79) | 372 (33) | 668 (37)
Statistical Analysis 1: Comparison: Aromatase Inhibitor vs Growth Hormone vs Aromatase Inhibitor and Growth Hormone; Test type: Superiority; p < 0.0001, ANOVA

8. Secondary Outcome: Change in Estradiol
Description: Those taking AI alone or AI/GH combined were grouped by type, either anastrozole or letrozole.
Time Frame: 0 to 24 months
Population: Of the 51 AI alone or AI/GH combined Subjects, 41 completed all procedures at 24 months, however, 1 Subject did not have Estrone results available for the 24 month visit (N=40).
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Anastrozole: Anastrozole 1mg for 2 to 3 years .
- Letrozole: Letrozole 2.5mg daily orally for 2 to 3 years .
Arm/Group | Anastrozole | Letrozole
Number analyzed (Participants) | 18 | 22
pg/mL | 8 (1) | 4 (1)
Statistical Analysis 1: Comparison: Anastrozole vs Letrozole; Test type: Superiority; p = 0.0003, ANCOVA

9. Secondary Outcome: Change in Estrone
Time Frame: 0 to 24 months
Population: Of the 76 Subjects, 65 completed all procedures at 24 months, however, 1 Subject, did not have Estrone results available for the 24 month visit (N=64).
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
Number analyzed (Participants) | 18 | 24 | 22
pg/mL | 0.0 (1.7) | 6.1 (0.9) | -0.9 (1.3)

ADVERSE EVENTS:
Arm/Group | Aromatase Inhibitor | Growth Hormone | Aromatase Inhibitor and Growth Hormone
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 4/25 | 2/25 | 2/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatase Inhibitor (N=25) | Growth Hormone (N=25) | Aromatase Inhibitor and Growth Hormone (N=26)
Slipped capital femoral epiphysis (SCFE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Self Injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular Torsion (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tibial Fracture and Torn Meniscus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No